CLINICAL TRIAL: NCT00152919
Title: A Comparison of 2 Schedules of Meloxicam to Reduce Prostate Swelling in Permanent Seed Prostate Brachytherapy - A Randomized Phase III Trial
Brief Title: Mobicox: Study of Meloxicam to Reduce Prostate Swelling in Permanent Seed Prostate Brachytherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 03-0840-C
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Meloxicam

INTERVENTIONS:
Drug: Meloxicam

SUMMARY:
Swelling of the prostate can occur during and after a brachytherapy. This swelling can cause urinary problems ranging from difficulty voiding to urinary retention. The purpose of this study is to investigate whether Mobicox started one week before brachytherapy and then continued afterwards is more effective in reducing the risk of needing a catheter than Mobicox given only afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to receive prostate brachytherapy as per the Ontario Provincial Guidelines will be eligible for this study (i.e. prostate specific antigen [PSA] < 10, Gleason score <7, Stage <= T2a)

Exclusion Criteria:

* Patients already taking anti-inflammatory drugs
* Patients with allergic-type reactions, including asthma and urticaria, to aspirin or nonsteroidal anti-inflammatory agents (see product information)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To compare 2 schedules of MeloxicamTM given in the peri-operative period to reduce prostate swelling after permanent seed implantation for prostate cancer

SECONDARY OUTCOMES:
To determine the influence of different timing of MeloxicamTM administration on urinary toxicity and biochemical response after permanent seed implantation for prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Crook, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Crook J, Patil N, Wallace K, Borg J, Zhou D, Ma C, Pond G. A phase III randomized trial of the timing of meloxicam with iodine-125 prostate brachytherapy. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):496-501. doi: 10.1016/j.ijrobp.2009.04.078. Epub 2010 Mar 28. PMID 20350785